CLINICAL TRIAL: NCT05584228
Title: SyMptomAtic Stricturing Small Bowel CRohn's Disease - Medical Treatment Versus Surgery, a Prospective, Multi-centre, Randomized, Non-inferiority Trial
Brief Title: Medical Treatment Versus Surgery in Stricturing Small Bowel Crohn's Disease
Acronym: SMART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC22_0408
Record Dates: First submitted 2022-09-26; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Crohn Disease
Keywords: Crohn's disease; stricture; resection; infliximab; azathioprine
MeSH Terms: conditions — Crohn Disease; Constriction, Pathologic | interventions — Azathioprine; Infliximab; CT-P13

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical treatment (Experimental): Combination therapy with subcutaneous infliximab and azathioprine
  Interventions: Drug: Azathioprine + infliximab
- Surgery (Active Comparator): Intestinal resection
  Interventions: Procedure: Intestinal resection

INTERVENTIONS:
Drug: Azathioprine + infliximab — Combination therapy using 2-2.5 mg/kg oral azathioprine plus subcutaneous infliximab
  Other Names: Imurel, Remsima
  Arms: Medical treatment
Procedure: Intestinal resection — Ileocolonic or small bowel resection
  Arms: Surgery

SUMMARY:
The objective of the SMART trial is to compare a combination therapy using azathioprine and subcutaneous infliximab versus ileocecal resection in patients with symptomatic small bowel Crohn's disease.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic, disabling and destructive inflammatory bowel disease (IBD) leading to progressive and cumulative bowel damage, including fistulas and strictures. Strictures are defined as intestinal luminal narrowing and can lead to obstructive symptoms in the medium-to-long term. Symptomatic strictures significantly impair patient's quality of life by the presence of obstructive symptoms such as abdominal pain, nausea, vomiting, abdominal distension, and dietary restrictions leading to malnutrition. Strictures can appear anywhere in the gastrointestinal tract, but affect most commonly the terminal ileum. Epidemiological studies indicate that more than 40% of patients with ileal CD will develop strictures.

However, treatment strategies are not well-defined in this indication. Most patients undergo surgery but recent observations indicate that a medical treatment by anti-TNF may be considered in stricturing CD. The European Crohn's Colitis Organization recommends that "ileocecal CD with obstructive symptoms, but no significant evidence of active inflammation, should be treated by surgery". However, the lack of inflammation is difficult to demonstrate and does not predict the extent of fibrosis, and inflammation and fibrosis are often associated. Thus, there is a need for better defining therapeutic strategies.

The objective of the SMART trial is to compare for the first time medical versus surgical approaches in stricturing CD. Indeed, up to date, no randomized controlled trial has been conducted to compare medical treatment alone versus surgery in patients with symptomatic stricturing CD. The hypothesis is that medical treatment by a combination therapy using infliximab and azathioprine is non-inferior to surgical resection in terms of health-related quality of life (HRQoL) at 1 year, with the advantage of being conservative as regards the high rates of post-operative recurrence with the subsequent risk of small bowel syndrome, as well as highly more acceptable by patients, especially since infliximab is now available as a biosimilar in a subcutaneous formulation, which should also improve the cost-effectiveness of the medical strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Male or female
* Documented small bowel CD with intestinal stricture(s) identified on CT, MRI or endoscopy, AND responsible for obstructive symptoms
* CREOLE score > 2

Exclusion Criteria:

* Adults under guardianship, safeguard justice or trusteeship
* Pregnant or breastfeeding female
* Acute bowel obstruction requiring urgent surgical intervention
* Suspected or confirmed gastrointestinal perforation
* Concurrent active perianal sepsis
* Internal fistulizing disease in association with strictures
* Colonic stenosis and/or colonic active disease at screening endoscopy
* Contra-indication to surgery, general anesthesia, anti-TNF, thiopurines
* Use of corticosteroids (prednisolone > 20 mg daily or equivalent) within 4 weeks prior to visit V0
* Treatment with any biologics within 8 weeks before visit V0
* Presence of a stoma
* HIV/HCV/HBV infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
IBD (inflammatory bowel disease) - related quality of life | 12 months
  Mean total inflammatory bowel disease questionnaire (IBDQ - Inflammatory Bowel Disease Questionnaire ) score.
  The total score ranges from 32 to 224, the higher the score the better the quality of life.

SECONDARY OUTCOMES:
IBD (inflammatory bowel disease) -related quality of life | 1, 3, 6, 9, 18 and 24 months
  Mean total inflammatory bowel disease questionnaire (IBDQ - Inflammatory Bowel Disease Questionnaire ) score.
  The total score ranges from 32 to 224, the higher the score the better the quality of life.
Endoscopic remission | 6 months
  Proportion of patients achieving endoscopic remission at month 6 (SES-CD < 2 in case of medical treatment or Rutgeerts score < i,2 in case of resection)
Obstructive symptoms | 1, 3, 6, 9, 12, 18 and 24 months
  Mean total score of CDOS (CROHN'S DISEASE OBSTRUCTIVE SCORE ) Scale frome 0 to 6. 0 is the best outcome.
Clinical activity | 1, 3, 6, 9, 12, 18 and 24 months
  Mean total score of CDAI (CROHN'S DISEASE ACTIVITY INDEX ) Scale from 0 to 1100. 0 is the best outcome.
inflammatory biomarkers (fecal calprotectin) | 1, 6, 12, 18 and 24 months
  Mean values of fecal calprotectin
inflammatory biomarkers ( C-reactive protein [CRP]) | 1, 6, 12, 18 and 24 months
  Mean values of CRP
imaging parameters | 12 months
  Proportion of patients with an improvement in wall thickening, contrast enhancement, T2-signal increase, diffusion weighted-signal increase and length of pathological segment at month 12 as compared to screening imaging (MRI) by physician global assessment
treatment failures | 12 and 24 months
  Proportion of patients without any treatment failures
patient-reported outcomes (disability) | 1, 3, 6, 9, 12, 18 and 24 months
  Mean total score of IBD-DI (INFLAMMATORY BOWEL DISEASE DISABILITY INDEX ) Score from 0 to 100. 0 is the best outcome (no disability)
patient-reported outcomes (work productivity) | 1, 3, 6, 9, 12, 18 and 24 months
  Mean total score of WPAI (WORK PRODUCTIVITY AND ACTIVITY IMPAIRMENT QUESTIONNAIRE) In percentage from 0 to 100.
patient-reported outcomes (fatigue) | 1, 3, 6, 9, 12, 18 and 24 months
  Mean total score of FACIT-F (Functional Assessment of Chronic Illness Therapy ) scores from 0 to 52, with higher scores corresponding to less fatigue
patient-reported outcomes (body image) | 1, 3, 6, 9, 12, 18 and 24 months
  Mean total score of body image questionnaire Ranges from 0 to 30 and can be calculated by summing up the 10 items. A higher score means a higher level of body image disturbance
patient-reported outcomes (generic quality-of-life) | 1, 3, 6, 9, 12, 18 and 24 months
  Mean total score of SF-36 (QUESTIONNAIRE SHORT FORM 36 HEALTH SURVEY ) Score ranging from 0 to 100. A low score reflects a perception of poor health, loss of function, presence of pain. A high score reflects a perception of good health, absence of functional deficit and pain
patient-reported outcomes (anxiety/depression) | 1, 3, 6, 9, 12, 18 and 24 months
  Mean total score of HAD (Hospital Anxiety and Depression scale) 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus allowing two scores (maximum score for each score = 21). Minimum : 0. The best outcome is 0.
Patient's acceptability -patients refusing to be included | 24 months
  Number of screened patients refusing to be included
patient's acceptability - The reason | 24 months
  The reason for refusing
intervention-related adverse events | 24 months
  Proportion of patients with intervention (drug or surgery) -related adverse events during the study
efficiency of medical treatment compared to surgery as assessed by a cost-utility analysis performed from a collective perspective | 24 months
  Incremental cost-utility ratio (cost per Quality-Adjusted Life-Years, QALYs) from a collective perspective

IPD SHARING:
Plan to Share IPD: No